CLINICAL TRIAL: NCT05336175
Title: Biomarker Study: Heart Failure Patients at Risk for Vascular Dementia and Alzheimer's Disease Related Dementia [Supplement of: IND Enabling Studies for a Novel Mas Receptor Agonist for Treatment of Cognitive Impairment in Patients at Risk for Alzheimer's Disease Related Dementia]
Brief Title: Biomarker Study: Heart Failure Patients at Risk
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Lee Ryan, Professor and Department Head, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2106885512
Record Dates: First submitted 2022-02-16; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Heart Failure; Angiotensin(1-7)
MeSH Terms: conditions — Heart Failure | interventions — angiotensin I (1-7); Saline Solution

STUDY DESIGN:
Intervention Model Description: Following baseline assessments of cognitive function, MRI and plasma Nfl levels, 40 subjects who have consented to participate in the Ang-(1-7) sub-study and will be randomly assigned to be given either Ang-(1-7) (100 micrograms/kg/day via subcutaneous injection) for 90 days (n=30) or saline placebo (n=10).
Who Masked: Participant
Masking Description: Participants will not know which treatment they're receiving. Research staff and patients care providers will have access to which treatment patients are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ang-(1-7) (Experimental): 30 participants will take 100 micrograms of Ang-(1-7) a day via subcutaneous injection for 90 days
  Interventions: Drug: Angiotensin 1-7
- Saline Placebo (Placebo Comparator): 10 participants will take 100 micrograms of saline placebo a day via subcutaneous injection for 90 days
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Angiotensin 1-7 — A substance, Angiotensin-(1-7) [Ang-(1-7)], is known to decrease inflammation in the brain. This substance is naturally produced in the body and works by activating areas in the brain involved in memory. Previous studies examining the ability of Ang-(1-7) treatment to prevent memory loss post open-heart surgery found that 21 days of treatment with Ang-(1-7) protected memory post-surgery. Participants treated with Ang-(1-7) were protected from post-surgery increase in NfL levels. This clinical "sub-project" within the existing study will allow us to obtain preliminary data to evaluate the safety and efficacy of treatment with Ang-(1-7) to improve cognitive function and determine if this treatment is associated with changes in plasma levels of NfL protein.30 participants will take 100 micrograms of Ang-(1-7) per day via subcutaneous injection for 90 days.
  Arms: Ang-(1-7)
Drug: Saline solution — Saline solution will be given as a placebo intervention to 10 participants. These participants will take 100 micrograms of saline solution per day via subcutaneous injection for 90 days.
  Arms: Saline Placebo

SUMMARY:
In order to determine if NfL can be a prognostic biomarker for VCID, participants will undergo a baseline evaluation consisting of neuropsychological testing and a blood draw with a 12-month follow-up consisting of neuropsychological testing and blood draw. After indicated interest in the study, participants will be screened either in person during a regularly scheduled clinic visit or by phone for eligibility. After consenting, participants will be scheduled for a baseline testing session. One session, lasting about 3 hrs, will include neuropsychological testing and a blood draw. After completion of baseline testing, participants who agree to take part in the clinical trial will begin a 12-week treatment of Ang-(1-7) via daily subcutaneous injections. During the drug treatment, participants will be called weekly to ensure that everything is going well with the injections. After participants have completed the 12-week injection period, participants will be scheduled for a second appointment which will include a blood draw and neuropsychological testing. All participant will be scheduled for a 12-month follow-up, which will include a blood draw and neuropsychological testing. Participants will be called every second month by research staff for a brief update on changes to health status, and to increase compliance with the 12-month follow-up.

Our One-Year outcome for this study is to provide early proof-of-concept clinical trial data that will support a larger, more comprehensive NIH funded study on the safety and efficacy of Ang-(1-7) to prevent cognitive impairment in HF patients at risk for developing VCID/ADRD. Our Long-Term outcome is to demonstrate whether plasma NfL exhibits characteristics making it useful as a Prognostic Biomarker to predict cognitive decline in early heart disease-associated VCID and identify pre VCID-symptomatic in individuals with symptomatic HF. Our goal will be to use levels of plasma Nfl as an enrollment enrichment factor in future trials to allow enrollment or stratification of patients more likely to develop VCID or ADRD and be responsive to Ang-(1-7) therapy.

DETAILED DESCRIPTION:
The investigators are proposing that neurofilament light (NfL) polypeptide might serve as a prognostic biomarker in blood that can help predict clinical progression in early VCID and identify pre-VCID-symptomatic individuals with stage II-IV heart failure. Our ultimate goal will be to use levels of NfL in blood as an enrollment enrichment factor for clinical trial eligibility criterion to identify patients who are more likely to develop VCID/ADRD. This project will establish baseline and 12-month longitudinal NfL values in heart failure patients at risk for VCID and determine the association between absolute levels of NfL with measures of cognitive function in participants with stages II, III, and IV heart failure. The investigators will also determine whether baseline levels of NfL predict change in cognitive function over a 12 month period. Investigators will examine whether the substance Ang-(1-7) is safe and effective for improving cognitive impairment in heart failure patients. This project will establish if treatment with Ang-(1-7) modifies the absolute levels of plasma Nfl and the change in these values over 12- months.

Recruitment of eligible patients will be approached at the Banner University Medical Center-North Campus Clinic C after patients have been seen for a standard of care clinic visit. Patients being evaluated for heart failure will be seen at Sarver Heart Center. The heart failure patients' medical records may be pre-screened before being are contacted for participation in this project. The cardiologist or clinic staff will introduce the study to the patient and may present the flyer. If the patient indicates to the doctor or clinic staff that he/she would like to learn about the research study, with the participant's permission, the doctor or clinic staff will contact a member of the research staff, who will discuss or schedule a time to discuss participation in detail with the patient. Participants medical records will be accessed to determine cardiovascular health history.

If a patient is interested, trained study staff will go through the Informed Consent Form (ICF) with the patient in an available private room. During the study consent process, the purpose, procedures, and risks of the study will be explained. Each section of the consent form (attached) will be reviewed together with the participant. The researcher will solicit questions and allow ample time for answers. It will be made clear to potential participants that participation in this study is completely voluntary and participants care will not be affected by decisions regarding participation in this study. The participant will also be asked to sign an addendum to the consent form regarding sharing data with colleagues. A copy of the signed consent form will be given to each participant. Signed consent forms will be stored in a locked file cabinet in the lab and then stored in the Psychology Building. The estimated time for recruitment and consenting of subjects at this location will take 30-60 minutes allowing for a time of question/answers. Potential participants who would like more time, will be given an ICF to take home and review the aspects of the study. A visit will be scheduled to complete the consenting in person. Eligible participants may also be contacted by phone to discuss the study, but the ICF would be signed in person.

Participants will complete the medication training/"test out" procedures at the Sarver clinic with trained clinic staff. The Ang-(1-7) drug will be kept at a Banner Investigational Pharmacy.

Behavioral research will be conducted at the University of Arizona in the psychology building and/or at the Biosciences Research Laboratories (BSRL) Building. Data will be collected on computers using stimulus presentation software and using pen and paper and will take approximately 2 hours and will be analyzed using statistical software. Research assistants will be trained by the principal investigator to help with recruitment and consenting of study participants, conducting study procedures, and data coding and analyses.

Recruitment and Screening:

Patients being evaluated for heart failure will be seen at BUMC-North Campus Clinic C. The heart failure patients' medical records may be pre-screened before being contacted for participation in this project. The cardiologist or clinic staff will introduce the study to the patient and may present the flyer (attached). If the patient indicates to the doctor or clinic staff that he/she would like to learn about the research study, the doctor or clinic staff will contact a member of the research staff, who will discuss or schedule a time to discuss participation in detail with the patient. Participants medical records will be accessed to determine cardiovascular health history. After indicating interest in the study, participants will be screened for eligibility either in person during a regularly scheduled clinic visit or by phone. With the participant's permission, research personnel will contact the participant to complete the screening form (information that will be obtained includes age, sex, race/ethnicity, education, smoking status, cardiac disease status, and current medications, comorbidities such as diabetes mellitus, renal function, chronic lung disease, congestive heart failure, cerebrovascular disease, hypertension, history of Covid-19 (demographics form and Covid-19 questionnaire is attached). If the screening is conducted over the phone, before starting, participants will be read a disclosure statement (attached) assuring that all information given is confidential and will only be used to determine eligibility for participation.

Overview of Procedures:

Once screened, a baseline testing session will be scheduled lasting about 3 hours. The session lasting also approximately 3 hours will include cognitive testing and a blood draw. Questionnaires will also be given to the participants at both the initial visit and the 12-month follow-up visit which will take approximately a half hour to fill out. After completion of a baseline assessment, participants will be scheduled for a 12-month follow-up, which will include a blood draw and neuropsychological testing and will take approximately 2.5 hours. Participants will be called every second month by research staff for a brief update (approximately 10 minutes each, 50 minutes total)(script attached) on changes to health status and to increase compliance with the 12-month follow-up. Total approximate time commitment = 8 hours, 20 minutes.

Participants who are enrolled in the clinical trial will be scheduled for four appointments. A baseline testing session, a medication training session, a second cognitive testing and blood draw - following the 12-week injection period, and a 12-month follow-up.

Questionnaires will also be given to the participants at both the initial visit and the 12-month followup visit which will take approximately a half hour to fill out. After completion of a baseline assessment, participants will go to the

Sarver clinic to complete medication training and "test out" procedures, this will take approximately 2 hours. Participants will then begin a 12-week course of daily injections of Ang-(1-7). Participants will complete a second round of neuropsychological testing and another blood draw. Participants will be scheduled for a 12-month follow- up, which will include a blood draw and neuropsychological testing and will take approximately 2.5 hours. Participants will be called called weekly for the 12-week duration of injections and then every other month until the 12-month follow-up. These calls are to ensure that everything is going well with the injections and to increase compliance with the 12-month follow-up. During these calls, participants will be asked several questions regarding any updates or changes to health status (approximately 10 minutes each, 160 minutes total). Total approximate time commitment = 14hours and 40 minutes.

Blood draw. Participants will undergo the collection of whole blood via venipuncture blood draw. Blood draw procedures will be conducted by a phlebotomist at the University of Arizona. The phlebotomist will wear non-latex gloves, check that the participant is not allergic to alcohol, sterilize the skin using an alcohol prep pad, and dispose of all used sharps in a sharps disposal container. Blood will be preprocessed and stored in a -80 freezer. Blood draws will be used to obtain NfL levels, genetic data, for a PepSeq assay to measure viral peptides, to examine inflammatory biomarkers, to examine metabolic health markers, and other possible markers related to cognition and aging.

Neuropsychological testing. Tests will be administered at baseline, after the 12-week injection period, and at the 12 month follow-up. Each session will last approximately 2 hrs. The cognitive tests evaluate memory (verbal/visual associative memory, recognition, pattern separation), executive functions (updating/working memory, inhibition, switching), processing speed (simple, complex), and perceptual discrimination. Tests were chosen from the experimental cognitive aging literature to increase sensitivity to individual variability in normal aging. Memory tests (associative memory, pattern separation memory) are particularly sensitive to hippocampal functioning. Additional clinical neuropsychological tests will be administered including the MOCA, AVLT, and NAART, allowing us to compare our participants to existing cohorts such as the NACC and ADNI, and to evaluate the potential for preclinical dementia. (See attached file (NfL IRB Test and Questionnaire Descriptions.docx) for test stimuli and descriptions as well as the record sheets in TestMaterialsRecordSheets.pdf.) Some of these tests are given using pen and paper, others are on the computer. Participants will be given breaks during testing sessions as needed. The Patient Health Questionnaire-9 (PHQ-9; https://www.hrsa.gov/behavioral-health) will be administered to evaluate depression (attached in the Questionnaires.pdf document)

Surveys/Questionnaires. A packet of various questionnaires assessing lifestyle, sleep, and activities will be given to the participant at the baseline visit to either be filled out during the visit or be taken home between visits. This packet may include the Pittsburgh Sleep Quality Index, World Health Organization Disability Assessment Schedule 2.0, The World Health Organization Quality of Life Questionnaire, Rapid Assessment of Physical Activity, the Kansas City Cardiomyopathy Questionnaire, and the Instrumental Activities of Daily Living Survey. Investigators will also be giving a questionnaire about Covid-19. This questionnaire may be sent to participants via a link using an online form or given as a pen and paper questionnaire. The purpose of this questionnaire is gain insight on the participant's Covid-19 history and examine if there is a relationship to cognition. This questionnaire may be given to participants with the disclosure form before the consent process. The questionnaires will take about a half hour for each each visit.

Study Subcutaneous Injections (s.c.). Treatment will be administered by subcutaneous (under the skin) injection once a day in the lower abdomen, front or side of thigh, or upper arm for a course of 12-weeks. Participants will be given a treatment of either Ang-(1-7) or saline. Participants will be blind to medication assignment. These injections will need to be administered by participants or a caregiver after receiving audio and visual training. A "test-out" procedure demonstrating proficiency will be required. The "test-out" procedure will be discussed in detail with participants by the research staff. Subcutaneous injections are routinely self-administered at home by patients requiring therapies like insulin for the treatment of diabetes.

Participants will be asked to complete a daily treatment log(attached). The log will include when the study injection was completed each day. In addition, investigators will ask that participants record any differences in feeling or possible adverse events that the participant notices that may or may not be related to the study injections.

A courier service will be used to deliver the study drug, syringes, and treatment log to participant's home once every 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be included in the study if they are:

  * 45 years old and older
  * Diagnosed at least 90 days prior to enrollment with stable NYHA Class II-IV HF, with symptoms during mild or moderate exercise but not at rest (i.e., shortness of breath),
  * On a stable medical regimen and free from hospitalizations in the prior 30 days,
  * Fluent English speakers.

Exclusion Criteria:

* Participants will be excluded from the study if there is evidence of:

  * Decompensated heart failure
  * Symptoms or signs of active coronary ischemia
  * Systolic blood pressure <95 mmHg
  * Significant lung disease (FEV1< 1.5 L, pO2 <70 on room air, pCO2 >45)
  * Active substance abuse or a history of substance abuse with cocaine, ecstasy, LSD, or IV drugs
  * History of or current seizure disorder or on medications for seizures (with the exception of childhood febrile seizures)
  * Neurological, psychiatric, or medical illness or injury expected to interfere with cognitive function including but not limited to stroke, head injury, Alzheimer's, Parkinson's, or brain cancer
  * Current depression (Patient Health Questionnaire-9 score >10)
  * Any condition which may prevent the subject from adhering to the study protocol such as significantly impaired vision.\

Note: Participants that have contraindications for MRI may be enrolled, but will not take part in the MRI portion of the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Blood Biomarkers - Neurology 4-Pleax A, pTau-181, and pTau 231 as measured by the Quanterix Simoa Neurology 4-plex A and Simoa pTau-181 and 283 advantage kits | These measurements will be taken at baseline
  We will use the Quanterix Simoa Neurology 4-Plex A (N4PA) Advantage kit to measure Neurology 4-Plex A (GFAP, NF-light, Total Tau, UCH-L1 and the Simoa pTau-181 and 283 Advantage kits to measure pTau-181 and pTau 231.
Baseline evaluations of associative, verbal memory as measured by the verbal paired associates task (version 2) | These measurements will be taken at baseline
  The verbal paired associates task (version 2) will be used to evaluate associative, verbal memory. Scores can range from 0 to 36 with higher scores indicating better outcomes.
Baseline evaluations of associative, visual memory as measured by the Face Name Associative Memory Test | These measurements will be taken at baseline
  The Face Name Associative Memory Test will be used to evaluate associative, visual memory. Scores can range from 0 to 12 with higher scores indicating better outcomes.
Baseline evaluations of pattern separation memory as measured by the Mnemonic Similarity Task | These measurements will be taken at baseline
  The Mnemonic Similarity Task will be used to evaluate pattern separation memory. Scores can range from 0 to 1.0 with higher scores indicating better outcomes
Baseline evaluations of executive functions - updating/working memory as measured by the Keep Track Task | These measurements will be taken at baseline
  The Keep Track Task will be used to evaluate executive function - updating/working memory. Scores can range from 0 to 30 with higher scores indicating better performance.
Baseline evaluations of executive functions - switching as measured by the Number-Letter Task | These measurements will be taken at baseline
  The Number-Letter task will be used to evaluate executive function - switching. Scores can range from 0.2sec to 10 sec with higher scores indicating worse outcomes
Baseline evaluations of executive functions - attention/inhibition as measured by the Flanker Task | These measurements will be taken at baseline
  The Flanker Task will be used to evaluate executive function - attention/inhibition. Scores can range from 200ms - 2000ms with higher scores indicating worse outcomes
Baseline evaluations of processing speeds - simple/complex processing speeds as measured by the Deary-Liewald Reaction Time Task | These measurements will be taken at baseline
  The Deary-Liewald Reaction Time Task will evaluate processing speed - simple/complex processing speed. Scores can range from 200ms - 1500ms with higher scores indicating worse outcomes
Baseline evaluations of reading ability/vocabulary as measured by the North American Reading Test | These measurements will be taken at baseline
  The North American Reading Test will be used to evaluate reading ability/vocabulary. Scores can range from 0 to 61 with higher score indicating better outcomes
Baseline evaluations of global cognitive functioning as measured by the Montreal Cognitive Assessment | These measurements will be taken at baseline
  The Montreal Cognitive Assessment will be used to evaluate global cognitive functioning/ Scores can range from 0 - 30 with higher scores indicating better outcomes.
Participants sleep quality will be assessed as measured by the Pittsburgh Sleep Quality Index | These measurements will be taken at baseline
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. Scores can range from 0 to 21 with higher scores indicating worse outcomes
Participants quality of life will be assessed as measured by the World Health Organization Quality of Life - BREF (WHOQOL-BREF) | These measurements will be taken at baseline
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) will be used to assess participant's quality of life. Score can range from 3 to 40 with higher scores indicating better outcomes
Participants disability due to health/mental health conditions will be assessed as measured by the World Health Organization Disability Assessment Schedule 2.0 | These measurements will be taken at baseline
  The World Health Organization Disability Assessment Schedule 2.0 will be used to assess participant's disability due to health/mental health conditions. Scores can range from 7 to 36 with higher scores indicating worse outcomes.
Participants physical activity will be assessed as measured by Rapid Assessment of Physical Activity | These measurements will be taken at baseline
  The Rapid Assessment of Physical Activity will be used to assess participant's physical activity. Scores can range from 1 to 10 with higher scores indicating better outcomes.
Participants heart failure health status will be assessed as measured by the Kansas City Cardiomyopathy Questionnaire | These measurements will be taken at baseline
  The Kansas City Cardiomyopathy Questionnaire. Scores can range from 12 to 118 with higher scores indicating better outcomes
Participants independent living skills will be assessed as measured by the Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L) | These measurements will be taken at baseline
  The Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L). Scores can range from 0 to 8 with higher scores indicating better outcomes.
12-week Blood Biomarkers - Neurology 4-Pleax A, pTau-181, and pTau 231 as measured by the Quanterix Simoa Neurology 4-plex A and Simoa pTau-181 and 283 advantage kits | These measurements will be taken after the 12 week drug course
  We will use the Quanterix Simoa Neurology 4-Plex A (N4PA) Advantage kit to measure Neurology 4-Plex A (GFAP, NF-light, Total Tau, UCH-L1 and the Simoa pTau-181 and 283 Advantage kits to measure pTau-181 and pTau 231.
12-week evaluations of associative, verbal memory as measured by the verbal paired associates task (version 2) | These measurements will be taken after the 12 week drug course
  The verbal paired associates task (version 2) will be used to evaluate associative, verbal memory. Scores can range from 0 to 36 with higher scores indicating better outcomes.
12-week evaluations of associative, visual memory as measured by the Face Name Associative Memory Test | These measurements will be taken after the 12 week drug course
  The Face Name Associative Memory Test will be used to evaluate associative, visual memory. Scores can range from 0 to 12 with higher scores indicating better outcomes.
12-week evaluations of pattern separation memory as measured by the Mnemonic Similarity Task | These measurements will be taken after the 12 week drug course
  The Mnemonic Similarity Task will be used to evaluate pattern separation memory. Scores can range from 0 to 1.0 with higher scores indicating better outcomes
12-week evaluations of executive functions - updating/working memory as measured by the Keep Track Task | These measurements will be taken after the 12 week drug course
  The Keep Track Task will be used to evaluate executive function - updating/working memory. Scores can range from 0 to 30 with higher scores indicating better performance.
12-week evaluations of executive functions - switching as measured by the Number-Letter Task | These measurements will be taken after the 12 week drug course
  The Number-Letter task will be used to evaluate executive function - switching. Scores can range from 0.2sec to 10 sec with higher scores indicating worse outcomes
12-week evaluations of executive functions - attention/inhibition as measured by the Flanker Task | These measurements will be taken after the 12 week drug course
  The Flanker Task will be used to evaluate executive function - attention/inhibition. Scores can range from 200ms - 2000ms with higher scores indicating worse outcomes
12-week evaluations of processing speeds - simple/complex processing speeds as measured by the Deary-Liewald Reaction Time Task | These measurements will be taken after the 12 week drug course
  The Deary-Liewald Reaction Time Task will evaluate processing speed - simple/complex processing speed. Scores can range from 200ms - 1500ms with higher scores indicating worse outcomes
12-week evaluations of reading ability/vocabulary as measured by the North American Reading Test | These measurements will be taken after the 12 week drug course
  The North American Reading Test will be used to evaluate reading ability/vocabulary. Scores can range from 0 to 61 with higher score indicating better outcomes
12-week evaluations of global cognitive functioning as measured by the Montreal Cognitive Assessment | These measurements will be taken after the 12 week drug course
  The Montreal Cognitive Assessment will be used to evaluate global cognitive functioning/ Scores can range from 0 - 30 with higher scores indicating better outcomes.
12-month Blood Biomarkers - Neurology 4-Pleax A, pTau-181, and pTau 231 as measured by the Quanterix Simoa Neurology 4-plex A and Simoa pTau-181 and 283 advantage kits | These measurements will be taken at the 12 month follow up
  We will use the Quanterix Simoa Neurology 4-Plex A (N4PA) Advantage kit to measure Neurology 4-Plex A (GFAP, NF-light, Total Tau, UCH-L1 and the Simoa pTau-181 and 283 Advantage kits to measure pTau-181 and pTau 231.
12-month evaluations of associative, verbal memory as measured by the verbal paired associates task (version 2) | These measurements will be taken at the 12 month follow up
  The verbal paired associates task (version 2) will be used to evaluate associative, verbal memory. Scores can range from 0 to 36 with higher scores indicating better outcomes.
12-month evaluations of associative, visual memory as measured by the Face Name Associative Memory Test | These measurements will be taken at the 12 month follow up
  The Face Name Associative Memory Test will be used to evaluate associative, visual memory. Scores can range from 0 to 12 with higher scores indicating better outcomes.
12-month evaluations of pattern separation memory as measured by the Mnemonic Similarity Task | These measurements will be taken at the 12 month follow up
  The Mnemonic Similarity Task will be used to evaluate pattern separation memory. Scores can range from 0 to 1.0 with higher scores indicating better outcomes
12-month evaluations of executive functions - updating/working memory as measured by the Keep Track Task | These measurements will be taken at the 12 month follow up
  The Keep Track Task will be used to evaluate executive function - updating/working memory. Scores can range from 0 to 30 with higher scores indicating better performance.
12-month evaluations of executive functions - switching as measured by the Number-Letter Task | These measurements will be taken at the 12 month follow up
  The Number-Letter task will be used to evaluate executive function - switching. Scores can range from 0.2sec to 10 sec with higher scores indicating worse outcomes
12-month evaluations of executive functions - attention/inhibition as measured by the Flanker Task | These measurements will be taken at the 12 month follow up
  The Flanker Task will be used to evaluate executive function - attention/inhibition. Scores can range from 200ms - 2000ms with higher scores indicating worse outcomes
12-month evaluations of processing speeds - simple/complex processing speeds as measured by the Deary-Liewald Reaction Time Task | These measurements will be taken at the 12 month follow up
  The Deary-Liewald Reaction Time Task will evaluate processing speed - simple/complex processing speed. Scores can range from 200ms - 1500ms with higher scores indicating worse outcomes
12-month evaluations of reading ability/vocabulary as measured by the North American Reading Test | These measurements will be taken at the 12 month follow up
  The North American Reading Test will be used to evaluate reading ability/vocabulary. Scores can range from 0 to 61 with higher score indicating better outcomes
12-month evaluations of global cognitive functioning as measured by the Montreal Cognitive Assessment | These measurements will be taken at the 12 month follow up
  The Montreal Cognitive Assessment will be used to evaluate global cognitive functioning/ Scores can range from 0 - 30 with higher scores indicating better outcomes.
Participants sleep quality will be assessed as measured by the Pittsburgh Sleep Quality Index | These measurements will be taken at the 12 month follow up
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. Scores can range from 0 to 21 with higher scores indicating worse outcomes
Participants disability due to health/mental health conditions will be assessed as measured by the World Health Organization Disability Assessment Schedule 2.0 | These measurements will be taken at the 12 month follow up
  The World Health Organization Disability Assessment Schedule 2.0 will be used to assess participant's disability due to health/mental health conditions. Scores can range from 7 to 36 with higher scores indicating worse outcomes.
Participants quality of life will be assessed as measured by the World Health Organization Quality of Life - BREF (WHOQOL-BREF) | These measurements will be taken at the 12 month follow up
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) will be used to assess participant's quality of life. Score can range from 3 to 40 with higher scores indicating better outcomes
Participants physical activity will be assessed as measured by Rapid Assessment of Physical Activity | These measurements will be taken at the 12 month follow up
  The Rapid Assessment of Physical Activity will be used to assess participant's physical activity. Scores can range from 1 to 10 with higher scores indicating better outcomes.
Participants heart failure health status will be assessed as measured by the Kansas City Cardiomyopathy Questionnaire | These measurements will be taken at the 12 month follow up
  The Kansas City Cardiomyopathy Questionnaire. Scores can range from 12 to 118 with higher scores indicating better outcomes
Participants independent living skills will be assessed as measured by the Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L) | These measurements will be taken at the 12 month follow up
  The Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L). Scores can range from 0 to 8 with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ryan, Ph.D., Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Banner - University Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No